CLINICAL TRIAL: NCT07363512
Title: Efficacy and Safety of Radiotherapy Combined With Tislelizumab and Anlotinib in the Treatment of Hepatocellular Carcinoma Complicated With Portal Vein Tumor Thrombus
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, zhoujinxue,MD, Deputy Director of Hepatopancreatobiliary Surgery Department, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-588-001
Record Dates: First submitted 2026-01-03; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: HCC - Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — tislelizumab; anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radiotherapy combined with tislelizumab and anlotinib (Experimental)
  Interventions: Combination Product: Radiotherapy combined with tislelizumab and anlotinib

INTERVENTIONS:
Combination Product: Radiotherapy combined with tislelizumab and anlotinib — Radiotherapy was performed using conventional fractionation. The PTV of the primary tumor and portal vein tumor thrombus was DT45-50Gy/25f, and the GTV was simultaneously pushed at DT50-60Gy/25f， Tislelizumab 200mg IV Q3W Anlotinib 12MG PO QD for two weeks followed by a one-week break Q3W

SUMMARY:
For HCC patients with PVTT who the researchers believe can benefit from radiotherapy combined with tislelizumab and anlotinib, informed consent forms will be signed, and then they will receive the study treatment and be followed up. The research design is as follows:

First, radiotherapy was administered. Three days ±1 day after the start of radiotherapy, tislelizumab and anlotinib treatment were initiated. Each cycle was three weeks, and the treatment continued until no toxicity was acceptable or clinical benefits were lost (evaluated by the researcher based on imaging, biochemical indicators, and the patient's clinical status).

ELIGIBILITY:
Inclusion Criteria:

1. Men aged between 18 and 75 or non-pregnant women;
2. Sign the informed consent form;
3. The researchers believe that the patients have the ability to comply with the research protocol;
4. Hepatocellular carcinoma (HCC) is diagnosed histologically, cytologically or clinically. Patients with liver cirrhosis are clinically diagnosed according to the AASLD standard, while non-liver cirrhosis patients need to be confirmed by histology.
5. Imaging examinations confirmed the presence of portal vein tumor thrombus;
6. The disease is not suitable for radical surgery;
7. Has not received any anti-tumor treatment in the past;
8. At least one measurable (measurable according to RECIST1.1) untreated lesion;
9. Tumor tissue samples before treatment (if available). If tumor tissue is available, submit one formalin-fixed, paraffin-embedded (FFPE) tumor sample in a paraffin block (preferred), or approximately 10-15 slides containing unstained, freshly cut, series sections, along with a relevant pathological report within 4 weeks of enrollment. If the FFPE samples described above are not available, any type of sample (including fine needle aspiration biopsy samples and cell mass samples) can also be accepted. A relevant pathological report should be provided along with the sample.
10. The ECOG performance status score is 0 or 1;
11. Child-Pugh grade A;
12. Adequate hematology and organ function, based on the following laboratory test results obtained within 7 days before enrollment (unless otherwise specified) : absolute neutrophil count (ANC)≥1.5×109/L (1500/μL), no granulocyte colony-stimulating factor support; Lymphocyte count ≥0.5×109/L (500/μL); Platelet count ≥50×109/L (50,000 /μL), no blood transfusion; Hemoglobin ≥90 g/L (9g/dL);
13. Before enrollment, any acute and clinically significant treatment-related toxicity (caused by previous treatment) must have been alleviated to ≤ grade 1, except for alopecia.
14. The result of the HIV antibody test during screening was negative;
15. Patients with active hepatitis B virus (HBV) infection: HBV DNA obtained within 28 days before randomization < 2000IU/mL, and having received at least 14 days of anti-HBV treatment (treated according to local standard treatment, such as entecavir) before randomization and willing to continue treatment during the study period.

Exclusion Criteria:

1. Current or previous history of autoimmune diseases or immune deficiencies
2. History of meningitis;
3. Idiopathic pulmonary fibrosis, organizing pneumonia (e.g., obliterative bronchiolitis), drug-induced pneumonia or idiopathic pneumonia, or evidence of active pneumonia can be seen on chest computed tomography (CT) images during the screening period. Radiation pneumonia has been allowed in the radiation area (fibrosis).
4. Known active tuberculosis;
5. Having major cardiovascular diseases (such as New York Heart Society Class II or more severe heart disease, myocardial infarction or cerebrovascular accident), unstable arrhythmia or unstable angina pectoris within 3 months prior to enrollment;
6. History of congenital long QT syndrome or corrected QT interval at screening >500ms (calculated using the Fridericia method);
7. A history of uncorrectable electrolyte disorders such as serum potassium, calcium or magnesium;
8. Received major surgical treatment (excluding diagnosis) within 4 weeks before enrollment or is expected to require major surgical treatment during the study period;
9. Malignant tumors other than HCC that have occurred within 5 years prior to enrollment, excluding those with negligible risk of metastasis or death (e.g., 5-year OS rate > 90%), such as well-treated cervical cancer in situ, non-melanoma skin cancer, localized prostate cancer, carcinoma in situ or stage I uterine cancer;
10. There was a severe infection within 4 weeks before enrollment, including but not limited to hospitalization due to infection, bacteremia or severe pneumonia complications;
11. Previous allogeneic stem cell or solid organ transplantation;
12. The patient cannot be followed up or is currently participating in other clinical trials;
13. Subjects who the researchers considered unsuitable for inclusion in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | The time from the start of the first medication to the occurrence of tumor shrinkage or disappearance and maintaining it for more than 4 weeks (up to 36 months).
  The proportion of patients whose tumor volume has shrunk by more than 20% and can be maintained for more than 4 weeks.

SECONDARY OUTCOMES:
Overall Survival | up to 36 months
Progression-Free Survival | up to 36 months
Disease Control Rate | up to 36 months
  The percentage of patients whose tumors shrank or remained stable over a period of time.
Duration of response | up to 36 months
Surgical resection rate | up to 36 months
  After the treatment of portal vein tumor thrombus downstaging, the researchers evaluated that surgical resection was feasible, which was considered a successful transformation. The proportion of those who ultimately underwent resection was the conversion rate of surgical resection.
adverse event | From the first treatment to 30 days after the end of the study
  Any adverse medical event that occurs to a patient or clinical trial subject after receiving a certain drug, but it does not necessarily have a causal relationship with the treatment.